CLINICAL TRIAL: NCT03443869
Title: A Phase III, Randomized, Double-Blind, Active Comparator-Controlled Study to Evaluate the Efficacy and Safety of MK-8228 (Letermovir) Versus Valganciclovir for the Prevention of Human Cytomegalovirus (CMV) Disease in Adult Kidney Transplant Recipients
Brief Title: Letermovir Versus Valganciclovir to Prevent Human Cytomegalovirus Disease in Kidney Transplant Recipients (MK-8228-002)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 8228-002; MK-8228-002 (Other: Merck); 2017-001055-30 (EudraCT Number)
Record Dates: First submitted 2018-02-19; First posted 2018-02-23 (Actual); Results first posted 2023-04-14 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: CMV Disease
MeSH Terms: interventions — letermovir; Valganciclovir; Acyclovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Letermovir (Experimental): LET 480mg (or 240 mg when administered concomitantly with cyclosporin A) tablet orally; placebo to VGCV tablet orally once daily; and 400 mg capsule of acyclovir (ACV) orally every 12 hours for 28 weeks
  Interventions: Drug: Letermovir; Drug: Acyclovir (ACV); Drug: Placebo to VGCV
- Valganciclovir (Active Comparator): 900 mg VGCV tablet orally, once daily; placebo to LET tablet orally once daily; and placebo to ACV orally every 12 hours for 28 weeks
  Interventions: Drug: Valganciclovir; Drug: Placebo to ACV; Drug: Placebo to LET

INTERVENTIONS:
Drug: Letermovir — LET 480mg (or 240 mg when administered concomitantly with cyclosporin A) once daily for 28 weeks
  Arms: Letermovir
Drug: Valganciclovir — 900 mg VGCV tablet orally, once daily for 28 weeks
  Arms: Valganciclovir
Drug: Acyclovir (ACV) — 400 mg over-encapsulated ACV tablet orally, every 12 hours for 28 weeks
  Arms: Letermovir
Drug: Placebo to ACV — Over-encapsulated placebo tablet orally, every 12 hours for 28 weeks
  Arms: Valganciclovir
Drug: Placebo to LET — Placebo to LET tablet orally, once daily for 28 weeks
  Arms: Valganciclovir
Drug: Placebo to VGCV — Placebo to VGCV tablet orally, once daily for 28 weeks
  Arms: Letermovir

SUMMARY:
The primary objective of this study is to evaluate the efficacy of letermovir (LET) versus valganciclovir (VGCV) in preventing CMV disease in adult kidney transplant recipients. The primary hypotheses are that LET is non-inferior to VGCV; and if non-inferiority is demonstrated, that LET is superior to VGCV, in preventing CMV disease through 52 weeks post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Have a documented negative serostatus for CMV within 180 days prior to randomization.
* Anticipate receiving a primary or secondary allograft kidney from a CMV IgG seropositive (D+) donor at the time of screening AND have received a primary or secondary allograft kidney from a documented D+ donor at the time of randomization.
* Be within 0 (i.e. day of transplantation) to 7 days (inclusive) post-kidney transplant at the time of randomization.
* Males agree to use contraception during the treatment period, and for at least 90 days after the last dose of study treatment, and refrain from donating sperm during this period.
* Female is not pregnant, not breastfeeding, and is not a woman of childbearing potential (WOCBP), OR if a WOCBP, agrees to follow the contraception guidance during the treatment period and for at least 90 days after the last dose of study treatment.

Exclusion Criteria:

* Has received a previous solid organ transplant or hematopoietic stem cell transplant (HSCT). Note: Participants who have received a prior primary allograft kidney may be enrolled, provided that all other inclusion/exclusion criteria are met.
* Is a multi-organ transplant recipient (e.g. kidney-pancreas). Double kidney transplant recipients (i.e. transplant of two kidneys from the same donor to the same recipient simultaneously) will be excluded.
* Has a history of CMV disease or suspected CMV disease within 6 months prior to randomization.
* Has suspected or known hypersensitivity to active or inactive ingredients of LET formulations, VGCV, GCV, and/or ACV formulations.
* Is on dialysis or plasmapheresis at the time of randomization. Dialysis includes hemofiltration.
* Has Child-Pugh Class C severe hepatic insufficiency at screening.
* Has both moderate hepatic insufficiency AND moderate-to-severe renal insufficiency at screening.
* Has any uncontrolled infection on the day of randomization.
* Has documented positive results for human immunodeficiency virus antibody (HIV-Ab) test at any time prior to randomization, or for hepatitis C virus antibody (HCV-Ab) and with detectable HCV ribonucleic acid (RNA) within 90 days prior to randomization, or hepatitis B surface antigen (HBsAg) within 90 days prior to randomization.
* Requires mechanical ventilation, or is hemodynamically unstable, at the time of randomization.
* Has a history of malignancy ≤5 years prior to signing informed consent.
* Is pregnant or expecting to conceive, is breastfeeding, or plans to breastfeed from the time of consent through at least 90 days following cessation of study therapy.
* Is expecting to donate eggs or sperm starting from the time of consent through at least 90 days following cessation of study therapy.
* Has received within 30 days prior to randomization or plans to receive during the study any of the following anti-CMV IgG antibody treatment or anti-CMV drug therapy including the following: Cidofovir, CMV hyper-immune globulin, Any investigational CMV antiviral agent/biologic therapy.
* Has received within 7 days prior to randomization or plans to receive during the study any of the following anti-CMV drug therapy: LET, GCV, VGCV, Foscarnet, ACV, Valacyclovir, Famciclovir.
* Is a user of recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence.
* Is currently participating or has participated in a study with an unapproved investigational compound or device within 28 days, or 5× half-life of the investigational compound whichever is longer, of initial dosing on this study.
* Has previously participated in this study or any other study involving LET.
* Has previously participated or is currently participating in any study involving administration of a CMV vaccine or another CMV investigational agent, or is planning to participate in a study of a CMV vaccine or another CMV investigational agent during the course of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 601 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (94):
- United States (27):
  - UAB ( Site 0269), Birmingham, Alabama
  - UCLA Medical Center ( Site 0266), Los Angeles, California
  - UC Davis Medical Center ( Site 0271), Sacramento, California
  - University of California-San Francisco ( Site 0236), San Francisco, California
  - Stanford Health Care ( Site 0235), Stanford, California
  - The Emory Clinic ( Site 0247), Atlanta, Georgia
  - University of Chicago ( Site 0251), Chicago, Illinois
  - Indiana University ( Site 0261), Indianapolis, Indiana
  - Ochsner Clinic Foundation ( Site 0238), New Orleans, Louisiana
  - University of Maryland Medical Center ( Site 0234), Baltimore, Maryland
  - Johns Hopkins Hospital ( Site 0232), Baltimore, Maryland
  - Brigham & Women's Hospital ( Site 0244), Boston, Massachusetts
  - Henry Ford Hospital ( Site 0242), Detroit, Michigan
  - University of Nebraska Medical Center ( Site 0272), Omaha, Nebraska
  - Saint Barnabas Medical Center ( Site 0250), Livingston, New Jersey
  - Icahn School of Medicine at Mount Sinai ( Site 0256), New York, New York
  - Columbia University Medical Center ( Site 0255), New York, New York
  - New York Presbyterian Hospital - Weill Cornell Medical Center ( Site 0276), New York, New York
  - Duke University Medical Center ( Site 0243), Durham, North Carolina
  - Wake Forest University Baptist Medical Center ( Site 0260), Winston-Salem, North Carolina
  - The Ohio State University Wexner Medical Center ( Site 0264), Columbus, Ohio
  - University of Pennsylvania ( Site 0270), Philadelphia, Pennsylvania
  - University of Pittsburgh ( Site 0252), Pittsburgh, Pennsylvania
  - Medical University of South Carolina ( Site 0257), Charleston, South Carolina
  - Vanderbilt University Medical Center ( Site 0275), Nashville, Tennessee
  - Virginia Commonwealth University ( Site 0245), Richmond, Virginia
  - University of Washington Medical Center ( Site 0246), Seattle, Washington
- Argentina (6):
  - Hospital El Cruce Nestor Carlos Kirchner ( Site 0351), San Juan Bautista, Buenos Aires
  - CEMIC ( Site 0352), Buenos Aires, Buenos Aires F.D.
  - Instituto de Nefrologia Nephrology S.A. ( Site 0182), Buenos Aires
  - Hospital Italiano de Buenos Aires ( Site 0188), CABA
  - Instituto de Cardiología de Corrientes Juana F. Cabral ( Site 0181), Corrientes
  - Clinica de nefrologia urologia y enfermedades cardiovasculares ( Site 0354), Santa Fe
- Australia (6):
  - Royal Prince Alfred Hospital ( Site 0005), Camperdown, New South Wales
  - Westmead Hospital ( Site 0006), Westmead, New South Wales
  - Princess Alexandra Hospital ( Site 0004), Woolloongabba, Queensland
  - Royal Adelaide Hospital ( Site 0003), Adelaide, South Australia
  - Monash Health-Monash Medical Centre ( Site 0008), Clayton, Victoria
  - Royal Melbourne Hospital ( Site 0007), Parkville, Victoria
- Austria (2):
  - Medizinische Universitat Innsbruck ( Site 0033), Innsbruck, Tyrol
  - Allgemeines Krankenhaus Universitaetskliniken Wien ( Site 0032), Vienna
- Belgium (3):
  - Universitair Ziekenhuis Antwerpen ( Site 0041), Edegem, Antwerpen
  - Cliniques Universitaires de Bruxelles - CUB - Hopital Erasme ( Site 0042), Brussels, Bruxelles-Capitale, Region de
  - UZ Leuven - Campus Gasthuisberg ( Site 0044), Leuven, Vlaams-Brabant
- Canada (5):
  - University of Alberta Hospital ( Site 0221), Edmonton, Alberta
  - Vancouver General Hospital ( Site 0224), Vancouver, British Columbia
  - St. Paul's Hospital ( Site 0225), Vancouver, British Columbia
  - Toronto General Hospital ( Site 0222), Toronto, Ontario
  - Hopital Maisonneuve-Rosemont CIUSSS de l Est de L Ile de Montreal ( Site 0226), Montreal, Quebec
- Colombia (8):
  - Hospital San Vicente Fundación - Rionegro ( Site 0205), Rionegro, Antioquia
  - Clinica del Country ( Site 0208), Bogotá, Bogota D.C.
  - Clinica Colsanitas S.A. Sede Clinica Universitaria Colombia ( Site 0209), Bogotá, Bogota D.C.
  - Hospital Universitario Mayor Mederi CIMED ( Site 0206), Bogotá, Bogota D.C.
  - Sociedad de Cirugia de Bogota Hospital de San Jose ( Site 0203), Bogotá, Bogota D.C.
  - Fundacion Cardiovascular de Colombia ( Site 0210), Bucaramanca, Santander Department
  - Fundacion Valle del Lili ( Site 0285), Cali, Valle del Cauca Department
  - Centro Medico Imbanaco de Cali S.A ( Site 0201), Cali, Valle del Cauca Department
- France (7):
  - Hopital Pasteur ( Site 0053), Nice, Alpes-Maritimes
  - CHU de Bordeaux. Hopital Pellegrin ( Site 0055), Bordeaux, Gironde
  - CHU Rangueil ( Site 0054), Toulouse, Haute-Garonne
  - C.H.R.U Bretonneau ( Site 0051), Tours, Indre-et-Loire
  - Hopital Henri Mondor du Creteil ( Site 0063), Créteil, Val-de-Marne
  - CHU - Hopital de Bicetre ( Site 0060), Le Kremlin-Bicêtre, Val-de-Marne
  - Hopital Tenon ( Site 0061), Paris
- Germany (3):
  - Medizinische Hochschule Hannover ( Site 0073), Hanover, Lower Saxony
  - Universitaetsklinikum Essen ( Site 0074), Essen, North Rhine-Westphalia
  - Charite Universitaetsmedizin Berlin ( Site 0071), Berlin
- Hungary (4):
  - Pecsi Tudomanyegyetem AOK ( Site 0282), Pécs, Baranya
  - Szegedi Tudomanyegyetem ( Site 0284), Szeged, Csongrád megye
  - Semmelweis Egyetem ( Site 0281), Budapest
  - Debreceni Egyetem. ( Site 0283), Debrecen
- Italy (4):
  - A.O.U. Citta della Salute e della Scienza di Torino ( Site 0096), Turin, Piedmont
  - Azienda Ospedaliera di Padova U.O.C. Trapianti Rene e Pancreas ( Site 0091), Padua, Veneto
  - IRCCS Ospedale San Raffaele di Milano ( Site 0098), Milan
  - Policlinico Gemelli Instituto di Clinica Chirurgica ( Site 0093), Roma
- Mexico (5):
  - Instituto Mexicano de Trasplantes S C ( Site 0212), Cuernavaca, Morelos
  - Centenario Hospital Miguel Hidalgo ( Site 0215), Aguascalientes
  - Instituto Nacional de Cardiologia Ignacio Chavez ( Site 0213), Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran ( Site 0214), Mexico City
  - Faicic S de RL de CV ( Site 0211), Veracruz
- Auckland City Hospital ( Site 0002), Auckland, New Zealand
- Poland (5):
  - Szpital Wojewodzki w Poznaniu ( Site 0168), Poznan, Greater Poland Voivodeship
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego ( Site 0162), Wroclaw, Lower Silesian Voivodeship
  - Szpital Kliniczny Dzieciatka Jezus ( Site 0165), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne ( Site 0170), Gdansk, Pomeranian Voivodeship
  - Pomorski Uniwersytet Medyczny ( Site 0167), Szczecin, West Pomeranian Voivodeship
- Spain (6):
  - Hospital del Mar ( Site 0121), Barcelona, La Coruna
  - Hospital Universitari de Bellvitge IDIBELL ( Site 0114), L'Hospitalet de Llobregat, La Coruna
  - Hospital Universitari Vall de Hebron ( Site 0112), Barcelona
  - Hospital Clinic i Provincial de Barcelona ( Site 0113), Barcelona
  - Hospital Doce de Octubre ( Site 0116), Madrid
  - Hospital Universitario Miguel Servet ( Site 0118), Zaragoza
- United Kingdom (2):
  - St Georges University Hospitals NHS Foundation Trust. ( Site 0136), London, London, City of
  - Queen Elizabeth Hospital ( Site 0356), Birmingham

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Limaye AP, Budde K, Humar A, Vincenti F, Kuypers DRJ, Carroll RP, Stauffer N, Murata Y, Strizki JM, Teal VL, Gilbert CL, Haber BA. Letermovir vs Valganciclovir for Prophylaxis of Cytomegalovirus in High-Risk Kidney Transplant Recipients: A Randomized Clinical Trial. JAMA. 2023 Jul 3;330(1):33-42. doi: 10.1001/jama.2023.9106. PMID 37279999
- [Derived] Strizki JM, Diamond TL, Teal VL, Gilbert CL, Wang W, Stauffer N, Haber BA. Cytomegalovirus Antiviral Resistance Among Kidney Transplant Recipients in a Phase 3 Trial of Letermovir vs Valganciclovir Prophylaxis. J Infect Dis. 2024 Dec 16;230(6):e1287-e1298. doi: 10.1093/infdis/jiae287. PMID 38853607
- [Derived] Vernooij RW, Michael M, Ladhani M, Webster AC, Strippoli GF, Craig JC, Hodson EM. Antiviral medications for preventing cytomegalovirus disease in solid organ transplant recipients. Cochrane Database Syst Rev. 2024 May 3;5(5):CD003774. doi: 10.1002/14651858.CD003774.pub5. PMID 38700045
- See also: Merck Clinical Trial Information — https://merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male/Female participants of at least 18 years of age with receipt of a kidney transplant were enrolled in this trial.
Groups:
- Letermovir: Letermovir (LET) 480 mg (or 240 mg when administered concomitantly with cyclosporin A) tablet orally; placebo to valganciclovir (VGCV) tablet orally once daily; and 400-mg capsule of acyclovir (ACV) orally every 12 hours for 28 weeks
Period: Overall Study
Arm/Group | Letermovir | Valganciclovir
Started | 301 | 300
Treated | 292 | 297
Completed | 256 | 266
Not Completed | 45 | 34
Not completed — Death | 3 | 3
Not completed — Withdrawal by Subject | 34 | 22
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 3 | 3
Not completed — Other | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Letermovir | Valganciclovir | Total
Number analyzed (Participants) | 301 | 300 | 601
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.6 (14.8) | 49.5 (15.1) | 49.6 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 90 | 174
  Male | 217 | 210 | 427
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56 | 45 | 101
  Not Hispanic or Latino | 230 | 240 | 470
  Unknown or Not Reported | 15 | 15 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 7
  Asian | 5 | 10 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 33 | 55
  White | 259 | 246 | 505
  More than one race | 9 | 6 | 15
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adjudicated Cytomegalovirus (CMV) Disease Through 52 Weeks Post-transplant
Description: CMV disease was defined as the presence of either CMV end-organ disease or CMV syndrome and was confirmed by an independent, blinded Clinical Adjudication Committee (CAC). Only CAC-confirmed ("adjudicated") cases were included in percentage of participants who met the endpoint. Investigator-assessed cases which were not confirmed by the CAC were not included.
Time Frame: Up to 52 weeks
Population: All randomized participants who received at least one dose of study treatment, were CMV seropositive organ donor/CMV seronegative organ recipient (D+/R-), and had no detectable CMV viral DNA (measured by central laboratory) on Day 1.
Measure: Number; unit: Percentage of Participants
Arm/Group | Letermovir | Valganciclovir
Number analyzed (Participants) | 289 | 297
Percentage of Participants | 10.4 | 11.8
Statistical Analysis 1: Comparison: Letermovir vs Valganciclovir; The Observed failure (OF) approach was used to handle missing values, that is participants who had discontinued prematurely from the study for any reason were not considered failures; Test type: Non-Inferiority — LET was concluded non-inferior to VGCV if the upper bound of the two-sided 95% CI for difference in percentage of participants with adjudicated CMV disease (LET - VGCV) was no higher than 10%; Stratum-adjusted Treatment Difference = -1.4, 95% CI 2-sided [-6.5 to 3.8] — Difference = LET minus VGCV

2. Secondary Outcome: Percentage of Participants With Adjudicated CMV Disease Through 28 Weeks Post-transplant
Description: CMV disease was defined as the presence of either CMV end-organ disease or CMV syndrome and was confirmed by an independent, blinded CAC. Only CAC-confirmed ("adjudicated") cases were included in percentage of participants who met the endpoint. Investigator-assessed cases which were not confirmed by the CAC were not included.
Time Frame: Up to 28 weeks
Population: All randomized participants who received at least one dose of study treatment, were D+/R-, and had no detectable CMV viral DNA (measured by central laboratory) on Day 1.
Measure: Number; unit: Percentage of Participants
Arm/Group | Letermovir | Valganciclovir
Number analyzed (Participants) | 289 | 297
Percentage of Participants | 0.0 | 1.7
Statistical Analysis 1: Comparison: Letermovir vs Valganciclovir; [analysis description as in outcome 1, analysis 1]; Test type: Other; Stratum-adjusted Treatment Difference = -1.7, 95% CI 2-sided [-3.4 to 0.1] — Difference = LET minus VGCV

3. Secondary Outcome: Time to Onset of Adjudicated CMV Disease Through 52 Weeks Post-transplant
Description: The time to onset of adjudicated CMV disease was calculated in days, from the day of randomization to the day of onset of CMV disease as determined by the CAC.
Time Frame: Up to 52 weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Letermovir | Valganciclovir
Number analyzed (Participants) | 289 | 297
Days | NA [NA to NA] — NA=The median time to event was not reached as fewer than half the participants reached this endpoint. | NA [NA to NA] — NA=The median time to event was not reached as fewer than half the participants reached this endpoint.

4. Secondary Outcome: Percentage of Participants With Any AE
Description: An AE was defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, was also an AE.
Time Frame: Up to 52 weeks
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Letermovir | Valganciclovir
Number analyzed (Participants) | 292 | 297
Percentage of Participants | 92.8 | 92.9
Statistical Analysis 1: Comparison: Letermovir vs Valganciclovir; Test type: Other; Difference in Percentages = -0.1, 95% CI 2-sided [-4.4 to 4.2] — Difference = LET minus VGCV

5. Secondary Outcome: Percentage of Participants With Any Drug-related Serious Adverse Event (SAE)
Description: An SAE was an AE that resulted in death, was life threatening, resulted in persistent or significant disability/incapacity, resulted in or prolonged an existing inpatient hospitalization, was a congenital anomaly/birth defect, was a cancer, was associated with an overdose, was another important medical event. SAEs that the investigator determined the relationship of the AE to the treatment as at least possibly related were reported.
Time Frame: Up to 52 weeks
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Letermovir | Valganciclovir
Number analyzed (Participants) | 292 | 297
Percentage of Participants | 1.4 | 5.1
Statistical Analysis 1: Comparison: Letermovir vs Valganciclovir; Test type: Other; Difference in Percentages = -3.7, 95% CI 2-sided [-7.0 to -0.9] — Difference = LET minus VGCV

ADVERSE EVENTS:
Time Frame: Up to 52 weeks
Description: All-Cause Mortality included all randomized participants. Non-serious and SAEs were reported for all randomized participants who received at least one dose of study treatment.
Groups:
- Letermovir: LET 480 mg (or 240 mg when administered concomitantly with cyclosporin A) tablet orally; placebo to VGCV tablet orally once daily; and 400-mg capsule of ACV orally every 12 hours for 28 weeks
Arm/Group | Letermovir | Valganciclovir
All-Cause Mortality (participants affected / at risk) | 5/301 | 3/300
Serious Adverse Events (participants affected / at risk) | 118/292 | 129/297
Other Adverse Events (participants affected / at risk) | 239/292 | 243/297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letermovir (N=292) | Valganciclovir (N=297)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 5 (5)
Hypoplastic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 9 (9)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (2) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 8 (8)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingivitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Overflow diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dehiscence (General disorders) | 1 (1) | 0 (0)
Discomfort (General disorders) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 1 (1) | 1 (1)
Implant site extravasation (General disorders) | 1 (1) | 0 (0)
Implant site necrosis (General disorders) | 1 (1) | 0 (0)
Malacoplakia (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Puncture site pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 9 (10) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 5 (5) | 3 (3)
Transplant rejection (Immune system disorders) | 6 (6) | 9 (9)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 1 (1)
Cytomegalovirus gastritis (Infections and infestations) | 2 (2) | 0 (0)
Cytomegalovirus hepatitis (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 7 (7) | 8 (8)
Cytomegalovirus syndrome (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus viraemia (Infections and infestations) | 2 (2) | 4 (5)
Endocarditis (Infections and infestations) | 1 (2) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Infected urinoma (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 3 (3)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0)
Lymph node tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Norovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Parvovirus B19 infection (Infections and infestations) | 1 (1) | 1 (1)
Parvovirus infection (Infections and infestations) | 1 (1) | 1 (1)
Penile gangrene (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia parainfluenzae viral (Infections and infestations) | 1 (1) | 0 (0)
Polyomavirus-associated nephropathy (Infections and infestations) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 4 (6) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1)
Renal graft infection (Infections and infestations) | 0 (0) | 2 (2)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Septic shock (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 8 (10) | 8 (10)
Urinary tract infection bacterial (Infections and infestations) | 1 (1) | 3 (4)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 1 (2)
Urosepsis (Infections and infestations) | 4 (5) | 4 (4)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Delayed graft function (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Graft complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Graft haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site erythema (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Post procedural urine leak (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Renal lymphocele (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Renal transplant failure (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Scapula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Transplant failure (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Urethral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Blood creatinine increased (Investigations) | 7 (7) | 3 (3)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 3 (4)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypervolaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
New onset diabetes after transplantation (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ocular lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Coma (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 8 (8) | 9 (12)
Bladder tamponade (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 1 (1)
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
IgA nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0)
Pyelocaliectasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal haematoma (Renal and urinary disorders) | 1 (1) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (1) | 3 (3)
Subcapsular renal haematoma (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 3 (3)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinoma (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 3 (3)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 3 (3)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 2 (2)
Iliac artery stenosis (Vascular disorders) | 1 (1) | 1 (1)
Lymphocele (Vascular disorders) | 8 (8) | 5 (5)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Letermovir (N=292) | Valganciclovir (N=297)
Anaemia (Blood and lymphatic system disorders) | 24 (25) | 34 (36)
Leukopenia (Blood and lymphatic system disorders) | 35 (46) | 105 (125)
Neutropenia (Blood and lymphatic system disorders) | 7 (9) | 50 (60)
Abdominal pain (Gastrointestinal disorders) | 21 (22) | 17 (17)
Constipation (Gastrointestinal disorders) | 27 (28) | 31 (36)
Diarrhoea (Gastrointestinal disorders) | 99 (130) | 85 (101)
Dyspepsia (Gastrointestinal disorders) | 19 (20) | 15 (17)
Nausea (Gastrointestinal disorders) | 35 (40) | 37 (48)
Vomiting (Gastrointestinal disorders) | 23 (31) | 26 (32)
Fatigue (General disorders) | 21 (21) | 34 (38)
Oedema peripheral (General disorders) | 44 (52) | 47 (61)
Pyrexia (General disorders) | 22 (24) | 24 (29)
Cytomegalovirus infection (Infections and infestations) | 8 (9) | 15 (15)
Polyomavirus viraemia (Infections and infestations) | 11 (11) | 16 (18)
Urinary tract infection (Infections and infestations) | 41 (51) | 45 (60)
Blood creatinine increased (Investigations) | 26 (29) | 39 (46)
White blood cell count decreased (Investigations) | 3 (4) | 15 (20)
Hyperglycaemia (Metabolism and nutrition disorders) | 10 (12) | 21 (22)
Hyperkalaemia (Metabolism and nutrition disorders) | 32 (36) | 38 (44)
Hypokalaemia (Metabolism and nutrition disorders) | 19 (22) | 10 (10)
Hypomagnesaemia (Metabolism and nutrition disorders) | 41 (44) | 40 (47)
Hypophosphataemia (Metabolism and nutrition disorders) | 35 (38) | 36 (41)
Back pain (Musculoskeletal and connective tissue disorders) | 18 (19) | 17 (18)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 (9) | 17 (19)
Dizziness (Nervous system disorders) | 15 (17) | 11 (14)
Headache (Nervous system disorders) | 23 (27) | 21 (27)
Tremor (Nervous system disorders) | 53 (56) | 52 (52)
Acute kidney injury (Renal and urinary disorders) | 15 (16) | 9 (10)
Dysuria (Renal and urinary disorders) | 16 (17) | 14 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 23 (26)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 22 (23)
Hypertension (Vascular disorders) | 38 (43) | 43 (46)
Hypotension (Vascular disorders) | 20 (21) | 13 (14)
Procedural pain (Injury, poisoning and procedural complications) | 8 (9) | 19 (22)
Metabolic acidosis (Metabolism and nutrition disorders) | 16 (17) | 14 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity was not directed by the sponsor, the investigator agreed to submit all manuscripts or abstracts to the sponsor before submission. This allowed the sponsor to protect proprietary information and to provide comments.

DOCUMENTS (2):
  • Study Protocol (2019-08-27): https://cdn.clinicaltrials.gov/large-docs/69/NCT03443869/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/69/NCT03443869/SAP_001.pdf